CLINICAL TRIAL: NCT01199237
Title: Effect of Anesthetic Choice (Sevoflurane Versus Desflurane) on Speed and Sustained Nature of Airway Reflex Recovery in the Context of Antagonized Neuromuscular Block
Brief Title: Impact of Anesthetic Choice (Sevoflurane Versus Desflurane) on Airway Reflex Recovery in the Context of Antagonized Neuromuscular Block
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H10722-35629-01
Record Dates: First submitted 2010-08-23; First posted 2010-09-10 (Estimated); Results first posted 2014-05-08 (Estimated); Last update posted 2014-05-16 (Estimated); Status verified 2014-05

CONDITIONS: Airway Reflexes, Protective; Recovery After Neuromuscular Block; Anesthetic Recovery
Keywords: Reflex, Pharyngeal; Anesthetics, Inhalation
MeSH Terms: conditions — Gagging; Respiratory Aspiration | interventions — Sevoflurane; Desflurane; Rocuronium; Neostigmine; Glycopyrrolate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sevoflurane (Active Comparator): Patients receive sevoflurane, rocuronium with neostigmine + glycopyrrolate reversal (70 and 14 ug/kg)
  Interventions: Drug: Sevoflurane; Drug: Rocuronium; Drug: Neostigmine; Drug: Glycopyrrolate
- Desflurane (Active Comparator): Patients receive Desflurane, rocuronium with neostigmine + glycopyrrolate reversal (70 and 14 ug/kg)
  Interventions: Drug: Desflurane; Drug: Rocuronium; Drug: Neostigmine; Drug: Glycopyrrolate

INTERVENTIONS:
Drug: Sevoflurane — Protective airway reflexes will be tested, judged by subject's ability to swallow 20 mL water
  Arms: Sevoflurane
Drug: Desflurane — Protective airway reflexes will be tested, judged by subject's ability to swallow 20 mL water
  Arms: Desflurane
Drug: Rocuronium
Drug: Neostigmine
Drug: Glycopyrrolate

SUMMARY:
Protective airway reflexes may be impaired in the postoperative period, creating the potential for aspiration of gastric contents, even after a patient exhibits appropriate response to command. Because assessment of airway reflex recovery is not possible in an intubated patient, the clinician must make an empiric decision as to when a patient is safe to extubate, and choose a combination of techniques least likely to result in pharyngeal impairment. Adequacy of reversal of neuromuscular block by cholinesterase inhibitors (e.g., neostigmine) is unpredictable, especially in the presence of profound paralysis, and tactile assessment of train-of four and sustained tetanus has shown poor correlation with objective assessments. Protective airway reflexes may also be impaired during early recovery by the anesthetics themselves, even when muscle relaxant has been avoided. In the absence of muscle relaxant the investigators previously demonstrated that patients receiving an anesthetic with higher tissue solubility, sevoflurane showed significantly greater impairment of swallowing up to 14 minutes after response to command compared to patients receiving an anesthetic with lower tissue solubility, desflurane. Therefore, we ask whether the combination of the more soluble anesthetic and the presence of neuromuscular block antagonized by neostigmine may create a multiplicative effect that might further prolong pharyngeal recovery. We plan to randomly assign 100 patients scheduled to undergo surgery with general anesthesia to a standardized anesthetic that includes 1) sevoflurane, rocuronium with 70 µg/kg neostigmine + 14 µg/kg glycopyrrolate antagonism (group S); or 2) desflurane, rocuronium with 70 µg/kg neostigmine + 14 µg/kg glycopyrrolate antagonism (group D). Airway reflex recovery will be judged as adequate by the patient's ability to swallow 20 mL of water without coughing or drooling 5, 10, 15, 20, 30 and 60 minutes after response to command. Anesthetic (sevoflurane or desflurane) will be discontinued after administration of reversal agent and recovery to TOF (train-of-four) ratio of 0.7.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1-2 patients
* Age 18-65 years
* body mass index (BMI) ≤ 35kg/m2
* Planned surgery requiring general anesthesia lasting approximately 1.5-3.0 hours
* Surgery requires or benefits from skeletal muscle relaxation
* All must pass the baseline 20 mL water swallowing test as previously described.

Exclusion Criteria:

* Pre-existing neuromuscular or central nervous system disorder
* Known condition interfering with gastric emptying
* Planned surgical procedure on the head or neck
* Known liver disease
* Serum creatinine > 1.5 mg/dL
* Concurrent use of neuroleptic medications
* Contraindication or previous adverse response to any of the study drugs
* Active asthma or reactive airways disease
* Surgery where upright position or brief cough would be contraindicated
* Inability to provide informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2010-08; Primary Completion 2012-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - UCSF Helen Diller Cancer Center, San Francisco, California
  - UCSF Moffitt-Long Hospital, San Francisco, California

REFERENCES:
- [Background] Sundman E, Witt H, Olsson R, Ekberg O, Kuylenstierna R, Eriksson LI. The incidence and mechanisms of pharyngeal and upper esophageal dysfunction in partially paralyzed humans: pharyngeal videoradiography and simultaneous manometry after atracurium. Anesthesiology. 2000 Apr;92(4):977-84. doi: 10.1097/00000542-200004000-00014. PMID 10754616
- [Background] Sundman E, Witt H, Sandin R, Kuylenstierna R, Boden K, Ekberg O, Eriksson LI. Pharyngeal function and airway protection during subhypnotic concentrations of propofol, isoflurane, and sevoflurane: volunteers examined by pharyngeal videoradiography and simultaneous manometry. Anesthesiology. 2001 Nov;95(5):1125-32. doi: 10.1097/00000542-200111000-00016. PMID 11684981
- [Background] Mckay RE, Large MJC, Balea MC, Mckay WR. Airway reflexes return more rapidly after desflurane anesthesia than after sevoflurane anesthesia. Anesth Analg. 2005 Mar;100(3):697-700. doi: 10.1213/01.ANE.0000146514.65070.AE. PMID 15728054
- [Background] McKay RE, Malhotra A, Cakmakkaya OS, Hall KT, McKay WR, Apfel CC. Effect of increased body mass index and anaesthetic duration on recovery of protective airway reflexes after sevoflurane vs desflurane. Br J Anaesth. 2010 Feb;104(2):175-82. doi: 10.1093/bja/aep374. Epub 2009 Dec 26. PMID 20037150
- [Background] Murphy GS, Szokol JW, Marymont JH, Greenberg SB, Avram MJ, Vender JS. Residual neuromuscular blockade and critical respiratory events in the postanesthesia care unit. Anesth Analg. 2008 Jul;107(1):130-7. doi: 10.1213/ane.0b013e31816d1268. PMID 18635478
- [Background] DePippo KL, Holas MA, Reding MJ. Validation of the 3-oz water swallow test for aspiration following stroke. Arch Neurol. 1992 Dec;49(12):1259-61. doi: 10.1001/archneur.1992.00530360057018. PMID 1449405

RESULTS

PARTICIPANT FLOW:
Recruitment Details: At one U.S. clinical site, patients scheduled to undergo surgery requiring general anesthesia lasting approximately 1.5 - 3.0 hours requiring tracheal intubation and paralysis during surgery were invited to participate
Pre-assignment Details: Participation of the first 26 enrollees was considered a pilot to determine the feasibility of measuring the primary outcome at T1+5 minutes. The majority of participants were alert, and no meaningful analyses could be made. The study was modified to assess the primary outcome at T1 + 2 minutes, and 81 additional participants were recruited.
Groups:
- Sevoflurane: Patients received sevoflurane, rocuronium with neostigmine + glycopyrrolate reversal (70 and 14 ug/kg)
- Desflurane: Patients received Desflurane, rocuronium with neostigmine + glycopyrrolate reversal (70 and 14 ug/kg)
Period: Overall Study
Arm/Group | Sevoflurane | Desflurane
Started | 41 | 40
Completed | 41 | 40
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sevoflurane | Desflurane | Total
Number analyzed (Participants) | 41 | 40 | 81
Age, Continuous [Mean (Full Range); unit: years] | 45.3 [42.0 to 48.7] | 43.3 [40.2 to 46.5] | 44.3 [40.2 to 48.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 36 | 77
  Male | 0 | 4 | 4
Region of Enrollment [Number; unit: participants]
  United States | 41 | 40 | 81

OUTCOME MEASURES:

1. Primary Outcome: Recovery of Ability to Swallow After Neostigmine/Glycopyrrolate Antagonism of Rocuronium Paralysis.
Description: The patient is judged by the primary anesthetist to be awake at time T1. At 2 minutes after T1, the patient was asked to swallow 20mL of water from a paper cup, and a blinded observer judged the ability to swallow based on transit of water to the posterior pharynx (absence of pooling or drooling) and absence of cough or gag.
Time Frame: At 2 minutes after response to command (T1).
Population: Only participants judged by the clinician as able to take the test (n=57)
Measure: Number; unit: participants
Arm/Group | Sevoflurane | Desflurane
Number analyzed (Participants) | 26 | 31
participants
  able to swallow at T1+2 minutes | 16 | 25
  unable to swallow at T1+2 minutes | 10 | 6
Statistical Analysis 1: Comparison: Sevoflurane vs Desflurane; Test type: Superiority or Other; p = 0.11, Chi-squared — Significant at p<0.05

2. Secondary Outcome: Time From Potent Inhaled Anesthetic Discontinuation to First Response to Command (T1)
Description: At the conclusion of surgery, after the patient's potent inhaled anesthetic was discontinued, the commands "open your eyes" and "squeeze my hand" were given at 30-second intervals. The time at which patient first appropriately response to both commands was noted as T1.
Time Frame: Up to 1 hour post-operative
Measure: Mean (Full Range); unit: seconds
Arm/Group | Sevoflurane | Desflurane
Number analyzed (Participants) | 41 | 40
seconds | 623 [509 to 736] | 343 [271 to 415]

3. Secondary Outcome: Nausea and Vomiting
Description: Patients were asked to rate their experience of nausea and vomiting on a 0-10 verbal analog scale, with 0 being absence and 10 being the worst imaginable
Time Frame: 30 minutes after T1
Population: Only participants able to respond at time of assessment
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Sevoflurane | Desflurane
Number analyzed (Participants) | 39 | 39
units on a scale
  Nausea | 0.385 [0 to 8] | 1.359 [0 to 8]
  Vomiting | 0 [0 to 0] | 0 [0 to 0]

4. Secondary Outcome: Nausea and Vomiting
Description: as for outcome 3
Time Frame: 60 minutes after T1
Population: Only patients able to respond at time of assessment
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Sevoflurane | Desflurane
Number analyzed (Participants) | 38 | 39
units on a scale
  Nausea | 0.263 [0 to 4] | 1.333 [0 to 10]
  Vomiting | 0 [0 to 0] | 0.026 [0 to 1]

5. Secondary Outcome: Time From Anesthetic Discontinuation to First Ability to Swallow
Description: At 2 minutes after first response to command (T1), the patient was asked to swallow 20 mL of water from a paper cup, and an observer blinded to anesthetic assignment assessed the ability to swallow based on transit of water to the posterior pharynx (absence of pooling or drooling) and absence of cough or gag (indicating misdirection of the water bolus into the laryngeal inlet). This test was repeated at 6, 14, 22, 30 and 60 minutes after the time of first response to command.
Time Frame: up to 60 minutes after T1
Measure: Mean (Full Range); unit: Seconds
Arm/Group | Sevoflurane | Desflurane
Number analyzed (Participants) | 41 | 40
Seconds | 1275 [947 to 1603] | 718 [513 to 922]

ADVERSE EVENTS:
Time Frame: 1-2 hours postoperatively
Arm/Group | Sevoflurane | Desflurane
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/40
Other Adverse Events (participants affected / at risk) | 0/41 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes